CLINICAL TRIAL: NCT01660698
Title: Immune-modulatory Effect of Candidate Probiotic Strain on Whole Blood Cells of Grass Pollen Allergic Individuals
Brief Title: Immune-modulatory Effect of Probiotic Strain on Grass Pollen Allergic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11.03.MET
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — maltodextrin; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): maltodextrin powder
  Interventions: Dietary Supplement: Maltodextrin
- Probiotic (Active Comparator): probiotic blended in maltodextrin
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Maltodextrin — maltodextrin powder
  Arms: Placebo
Dietary Supplement: Probiotic — probiotic blended in maltodextrin powder
  Arms: Probiotic

SUMMARY:
The purpose of the current study is to evaluate the effect of administering a probiotic strain on allergic symptoms and immune parameters (Th-2 cytokines, effector cells) in seasonal allergic rhinitis subjects.

DETAILED DESCRIPTION:
To identify immune markers in allergic individuals that are impacted by probiotic treatment during seasonal exposure

ELIGIBILITY:
Inclusion Criteria:

* Confirmed allergy (allergic rhinitis) to grass pollen > 1 year and positive SPT > 3mm wheal diameter to grass pollen.
* Age 20-65 years adults
* Body Mass Index 19- 29 (people in the normal and overweight range)
* Having obtained his/her informed consent.

Exclusion Criteria:

* Anemia
* Family history of congenital immunodeficiency
* Regular consumption of immunosuppressive or anti-inflammatory treatment
* Under medication against allergy (e.g. anti histaminic)
* Avoid regular consumption of probiotic and other dietary nutritional interventions
* Have a high alcohol consumption (more than 1 drink/day)
* Consumption of illicit drugs
* Pregnancy

  * Subject who cannot be expected to comply with the study procedures, including consuming the test products
  * Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Maurice Beaumont, MD, PhD, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- Metabolic Unit, Nestlé Research Center, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Singh A, Hacini-Rachinel F, Gosoniu ML, Bourdeau T, Holvoet S, Doucet-Ladeveze R, Beaumont M, Mercenier A, Nutten S. Immune-modulatory effect of probiotic Bifidobacterium lactis NCC2818 in individuals suffering from seasonal allergic rhinitis to grass pollen: an exploratory, randomized, placebo-controlled clinical trial. Eur J Clin Nutr. 2013 Feb;67(2):161-7. doi: 10.1038/ejcn.2012.197. Epub 2013 Jan 9. PMID 23299716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at the Metabolic Unit, (study no. 11.03.MET, NCT01660698) during the Grass Pollen (GP) season. Twenty seven adults volunteered, of which twenty four who gave written informed consent were screened for clinical history of allergy to GP > 2 years and a confirmatory skin prick test (SPT) to GP. Twenty subjects were randomized.
Pre-assignment Details: Subjects assigned to either: probiotic or placebo groups and taking assigned product for 8 weeks with three visits: V1(at baseline), V2 (4 weeks after treatment) and V3 (8 weeks after treatment).
Groups:
- Placebo: maltodextrin powder
  Maltodextrin : maltodextrin powder
- Probiotic: probiotic blended in maltodextrin
  Probiotic : probiotic blended in maltodextrin powder
Period: Overall Study
Arm/Group | Placebo | Probiotic
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Probiotic | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Inter-Quartile Range); unit: years] | 34 [29.25 to 44] | 35.5 [31.5 to 38] | 34.7 [29.25 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Th2 Cytokines (IL-13) Between Placebo and Probiotic Groups at Baseline (Beginning of Product Intake), 4 Weeks (Mid Period of Product Intake) and 8 Weeks (End of Product Intake)
Description: A maximum of 10 ml heparinized, venous blood will be collected during Visit 1, 2 and 3. Whole blood cells will be cultured for 120 hours (5 days) with culture medium with different stimuli. Cell supernatants will be collected and analyzed for different cytokines.
Time Frame: 0 (baseline), 1 and 2 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Probiotic
Number analyzed (Participants) | 10 | 10
ng/mL
  IL13 at V1 (beginning of product intake) | 1238 (1453) | 720 (854)
  IL13 at 1 month (4 weeks) | 975 (1019) | 998 (1383)
  IL13 at 2 months (8 weeks) | 968 (1206) | 218 (151)

2. Secondary Outcome: Comparison Between Probiotic and Placebo at Baseline (Beginning of Product Intake), 1 Month and 2 Months (End of Product Intake)
Description: TNSS Questionnaire were distributed at every visit (1 questionnaire for every week). The scored questionnaire were collected at subsequent visits. The symptom scores for nasal congestion, runny nose, nasal itching and sneezing were expressed as weekly sums (scale 0-3 for each symptom). The TNSS was the weekly sum for all the symptoms (scale 0-12). The TNSS data were analyzed as both monthly averages (at V2 and V3 compared to baseline V1) and weekly TNSS scores. Monthly TNSS scores were calculated as average over the 4 weeks preceding the visits. The higher the score is, the worse the outcome is.
Time Frame: Measures at baseline, 1, and 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Probiotic
Number analyzed (Participants) | 10 | 10
units on a scale
  TNSS score at baseline | 4.10 (3.11) | 4.90 (3.35)
  TNSS score at 1 month | 3.05 (1.86) | 3.92 (1.89)
  TNSS score at 2 months | 3.00 (2.04) | 1.50 (1.33)

3. Secondary Outcome: Change From Baseline in Pro-inflammatory Cytokines (TNF-alpha, IL-1beta) at 8 Weeks in ex Vivo Stimulated Whole Blood Cells
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Immunoglobulin Levels in Serum Between Treatment Groups
Time Frame: 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Basophil Activation at 8 Weeks in ex Vivo Stimulated Whole Blood Cells
Time Frame: 8 weeks
Reporting Status: Not Posted

6. Primary Outcome: Comparison of Th2 Cytokines (IL-5) Between Placebo and Probiotic Groups at Baseline (Beginning of Product Intake), 4 Weeks (Mid Period of Product Intake) and 8 Weeks (End of Product Intake)
Description: as for outcome 1
Time Frame: 0 (baseline), 1, and 2 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Probiotic
Number analyzed (Participants) | 10 | 10
ng/mL
  IL-5 at baseline (begining of product intake) | 1439 (1501) | 700 (683)
  IL-5 at 1 month (4 weeks) | 1191 (1005) | 980 (905)
  IL-5 at 2 months (8 weeks) | 1277 (956) | 323 (301)

ADVERSE EVENTS:
Time Frame: From baseline until 4 weeks following the last product intake
Description: All adverse events were documented on the the e-CRFs. In the case of a SAE persisting beyond trial termination, a follow up visit may be required. Any potential cause-effect relationship between the study product and the adverse event was assessed based on all examinations and laboratory analysis.
Arm/Group | Placebo | Probiotic
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No